CLINICAL TRIAL: NCT06621498
Title: Ridge Preservation Using Guided Regenaration, Platelet-rich Plasma and Free Gingival Grafts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Varna (Other)
Responsible Party: Principal Investigator, Ralitsa Yotsova, Dr., Medical University of Varna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 118/23.06.2022
Record Dates: First submitted 2024-09-27; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Post-Extraction Socket Healing; Ridge Preservation
Keywords: ridge preservation; post-extraction healing; post-extraction resorption; dense polytetrafluoroethylene membrane; free gingival graft; platelet-rich plasma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Ridge preservation with dense polytetrafluoroethylene membrane (Experimental): Tooth extraction and ridge prservation with dense PTFE membrane to cover the socket was used in this group.
  Interventions: Procedure: Ridge preservation technique
- Ridge preservation with dense polytetrafluoroethylene membrane and platelet-rich plasma (Experimental): Tooth extraction and ridge prservation with dense PTFE membrane and autologous PRP was used in this group.
  Interventions: Procedure: ridge preservation
- Ridge preservation with free gingival grafts (Experimental): Tooth extraction and ridge prservation with autologous free gingival grafts as a method for socket sealing was used. Donor sites were the hard palate and the maxillary tuberosity.
  Interventions: Procedure: ridge preservation
- Control group (No Intervention): Tooth extraction without ridge preservation.

INTERVENTIONS:
Procedure: Ridge preservation technique — Tooth extraction, deperiostation of the buccal and oral marginal gingiva, placement of d-PTFE membranes and suturing.
  Other Names: ridge preservation; socket preservation
  Arms: Ridge preservation with dense polytetrafluoroethylene membrane
Procedure: ridge preservation — Tooth extraction, socket filling with PRP, deperiostation of the buccal and oral marginal gingiva, placement of d-PTFE membranes and suturing.
  Other Names: socket preservation
  Arms: Ridge preservation with dense polytetrafluoroethylene membrane and platelet-rich plasma
Procedure: ridge preservation — Tooth extraction, full-thickness graft harversting and socket sealing with it.
  Other Names: socket preservation
  Arms: Ridge preservation with free gingival grafts

SUMMARY:
The goal of this clinical trial is to learn if ridge preservation methods with dense polytetrafluoroethylene membranes, with d-PTFE membranes and platelet-rich plasma, and with free gingival grafts can reduce vertical resorption of the post-extraction socket walls.

Researchers compared each experimental group to a control group (unassisted socket healing). Participants were randomly allocated to one of the four groups.

Cone-beam computed tomography was performed after the procedure and 3 months post-operatively to evaluate the vertical socket wall resorption.

ELIGIBILITY:
Inclusion Criteria:

1. Patients in the age group 18-65 years;
2. Patients in good general condition;
3. Patients requiring extraction of premolars or molars;
4. Patients in whom restoration of the missing tooth with a dental implant and/or prosthetic construction is planned;
5. Signed informed consent to participate in the study.

Exclusion Criteria:

1. Patients with contraindications for general surgical treatment:

   * patients with uncontrolled arterial hypertension;
   * patients with uncontrolled metabolic diseases;
   * patients with AMI in the last 6 months;
   * patients on hemodialysis treatment;
   * patients who underwent chemotherapy and/or radiotherapy in the last year;
   * patients on immunosuppressive therapy;
   * patients on anti-resorptive and anti-angiogenic therapy;
   * patients with concomitant acute diseases at the time of the study;
   * patients with proven psychiatric diseases;
   * pregnancy.
2. There are local contraindications:

   * insufficient volume of bone after the extraction to carry out RP;
   * acute inflammatory disease or tumor process in the area;
3. Lack of informed consent.
4. Lack of patient motivation for the treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-06-23 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-04-12 (Actual)

PRIMARY OUTCOMES:
Vertical post-extraction resorption of the socket walls | 3 months
  Each socket wall is measured using CBCT right after the extraction and after 3 months to assess the vertical resorption.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan V Peev, DsC, Principal Investigator — Medical University of Varna
Locations (1):
- Medical University Varna, Varna, Bulgaria

IPD SHARING:
Plan to Share IPD: No
It has not been approved by the Research Ethics Committee